CLINICAL TRIAL: NCT00108602
Title: Sleep Apnea: Mechanism and Cerebrovascular Consequences
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study of the overall grant was not pursued as the aims were changed
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Barczi, Steven - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: RESP-017-03S
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Sleep Apnea, Obstructive; Stroke
Keywords: sleep apnea; stroke; ventilatory control
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stroke; Sleep Apnea Syndromes | interventions — Acetazolamide

ARMS (1):
- 1 (Other)
  Interventions: Drug: acetazolamide

INTERVENTIONS:
Drug: acetazolamide

SUMMARY:
This study will determine the effect of ventilatory stimulation on obstructive sleep apnea in selected patients with stroke. We will select a subset of patients with stroke in the prior 3 months who are most likely to have ventilatory instability as a cause of the upper airway obstruction as indicated by the absence of obesity, an abnormal hypocapnic apnea threshold and resolution of obstructive apnea during CO2 administration. Following baseline polysomnography, patients will be randomly assigned to acetazolamide (250 mg hs [at bedtime]) versus placebo for 7 days. Polysomnography will be repeated and then subjects will cross-over therapies for another 7 days followed by a final nocturnal polysomnography.

DETAILED DESCRIPTION:
This study never enrolled patients. It was a component of a larger VA Merit grant and the other aims of the grant were completed but due to logistic issues and recruitment challenges this particular protocol was never made active.

ELIGIBILITY:
Inclusion Criteria:

* We will select non-obese patients (body mass index [BMI] <30 kg/m2) with stroke diagnosed during the 3 previous months and obstructive sleep apnea on screening sleep study (apnea-hypopnea index [AHI] >15 events/hr of study time).
* Patients with stroke will be selected based on the following criteria: 85 years old or less with a history of ischemic stroke within 3 months resulting in mild to moderate neurological impairment (Rankin scale < 3)

Exclusion Criteria:

* Hemorrhagic stroke,
* A history of chronic obstructive lung disease,
* Left ventricular ejection fraction (LVEF) <55%
* Evidence of nasal or pharyngeal obstruction on physical examination.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Barczi, MD, Principal Investigator — Wlliam S. Middleton Memorial Veterans Hospital, Madison